CLINICAL TRIAL: NCT05435352
Title: Prospective Evaluation of Image-based Artificial Intelligence Research and Development Tool for Precision Neoadjuvant Triple-Negative Breast Cancer Treatment
Brief Title: Image-based AI Predictive Biomarkers for Precision Neoadjuvant Triple-negative Breast Cancer Treatment
Acronym: PEAR-TNBC
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Ourotech, Inc. (Industry)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEAR-TNBC_ Protocol_v2.0
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer; Triple Negative Breast Neoplasms
Keywords: computer vision; cell culture; microtumor; functional testing; predictive biomarker
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Tumor cores
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early TNBC patient Cohort A: Early TNBC patients receiving neoadjuvant therapy and providing core needle biopsy.
  Any approved neoadjuvant therapy can be used based on physician's choice.
  Interventions: Procedure: Core needle biopsy
- Early TNBC patient Cohort B: Early TNBC patients receiving neoadjuvant therapy and providing core needle biopsy and blood.
  Any approved neoadjuvant therapy can be used based on physician's choice.
  Interventions: Procedure: Core needle biopsy

INTERVENTIONS:
Procedure: Core needle biopsy — An additional core needle biopsy is taken to run the Pear Bio test. Test results are not used to inform treatment. Approved neoadjuvant therapy regimens are given to the patient as per standard of care to observe response.

SUMMARY:
Pear Bio has developed an organ-on-a-chip device together with a computer vision pipeline through which the response of an individual patient's tumor to different chemotherapy regimens can be tested simultaneously ex vivo. This study will recruit patients with early TNBC who are planned for standard of care neoadjuvant chemotherapy followed by surgery. The oncologist will be blinded to the response on the Pear Bio tool (the assay will be run in parallel with the patient's neoadjuvant chemotherapy). The primary objective of this study is to establish the sensitivity and specificity of Pear Bio's test against patient outcomes (pathological complete response).

DETAILED DESCRIPTION:
This is a multicenter, UK-based, observational pilot study that aims to determine the accuracy of a new assay, the Pear Bio tool, in predicting pathological complete response (pCR) in patients receiving neoadjuvant chemotherapy for early TNBC. Patients will undergo an additional, mandatory biopsy of the breast tumor before commencing neoadjuvant chemotherapy. The biopsy sample will be run on the Pear Bio tool while the patient receives their standard of care neoadjuvant chemotherapy. As such, for this study, the result from the Pear Bio tool will not be used to inform the choice of neoadjuvant chemotherapy and the treating oncologist will be blinded to the assay results. The pathological outcome from surgery (pCR vs non-pCR) will be collected and used to calculate the specificity of the assay as the primary endpoint of the study. Sensitivity, positive predictive value and negative predictive value will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent prior to admission to this study.
* Female or male aged ≥18 years.
* Histologically confirmed invasive primary breast cancer which is triple-negative by the most recent ASCO/College of American Pathologists (CAP) guidelines.
* Stage I-III breast cancer planned for neoadjuvant chemotherapy followed by surgery.
* Primary breast tumor size ≥10 mm. For patients with bilateral tumors both of the breast tumors have to be TNBC and at least one has to be ≥10 mm.
* Willing to undergo a mandatory additional core needle biopsy from the primary breast mass prior to starting neoadjuvant chemotherapy. Patients with bilateral breast cancer only need to have one tumor biopsied if both tumors are ≥10 mm.
* Willing to donate 40mL of whole blood (cohort B only)

Exclusion Criteria:

* Inflammatory breast cancer.
* Inoperable or metastatic TNBC.
* Patients who have already commenced neoadjuvant chemotherapy.
* Treatment concurrently or within 4 weeks of commencing neoadjuvant chemotherapy with any experimental therapies. Patients who are due to receive standard of care neoadjuvant chemotherapy on the control arm of a trial may be eligible after discussion with the medical monitor.
* Secretory or adenoid cystic histological subtypes of triple-negative breast cancer.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early TNBC patients due to receive neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Pathological complete response correlation accuracy (specificity) | 6 months
  The specificity of Pear image-based biomarkers are established against patient pathological complete response (evaluated on surgical sample post-neoadjuvant therapy).

SECONDARY OUTCOMES:
Pathological complete response correlation accuracy (sensitivity) | 6 months
  The sensitivity of Pear image-based biomarkers are established against patient pathological complete response (evaluated on surgical sample post-neoadjuvant therapy).
Pathological complete response correlation accuracy (positive predictive value) | 6 months
  The positive predictive value of Pear image-based biomarkers are established against patient pathological complete response (evaluated on surgical sample post-neoadjuvant therapy).
Pathological complete response correlation accuracy (negative predictive value) | 6 months
  The negative predictive value of Pear image-based biomarkers are established against patient pathological complete response (evaluated on surgical sample post-neoadjuvant therapy).

OTHER OUTCOMES:
Culture success rate | 4 days
  The percentage of patient samples successfully arriving at central lab with >100k live cells isolated and maintaining 70% cell viability after 4 days in culture with no treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Manchester University NHS, Manchester

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data will be shared between study sites, such as treatment and outcome data for each patient. No publication will be made revealing individual patient data; only group-level data will be published.

REFERENCES:
- Available data/document: Study Protocol — https://www.pearbio.com/peartnbc